CLINICAL TRIAL: NCT05687708
Title: Effect of Non-nutritive Sucking Stimulation on Oral Intake and Early Feeding Skills in Newborns With Perinatal Asphyxia: A Randomized Controlled Trial
Brief Title: Effect of Non-nutritive Sucking on Transition to Oral Feeding in Infants With Asphyxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hilal Berber Çiftci, Doctoral Student, Speech and Language Therapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MedipolDKT
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Swallowing Disorder; Perinatal Asphyxia; Feeding; Difficult, Newborn; Feeding Disorder of Infancy or Early Childhood; Hypoxic-Ischemic Encephalopathy; Speech Therapy
Keywords: perinatal asphyxia; non-nutritive sucking; oral feeding; oral stimulation
MeSH Terms: conditions — Deglutition Disorders; Hypoxia-Ischemia, Brain; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Nutritive Sucking (Experimental): Non-Nutritive Sucking
  Interventions: Other: Non-Nutritive Sucking
- Control (No Intervention): routine treatment

INTERVENTIONS:
Other: Non-Nutritive Sucking — NNS is stimulated by giving stimulus into the baby's mouth with the help of a finger wearing gloves.
  Arms: Non-Nutritive Sucking

SUMMARY:
The transition period to full oral feeding in infants with perinatal asphyxia is important in predicting long-term outcomes. The transition to independent oral feeding is accepted as a discharge criterion by the American Academy of Pediatrics, and the long transition from tube feeding to oral feeding prolongs the discharge process. Prolonged transition to oral feeding increases maternal stress as it delays gastrointestinal problems, mother-infant interaction and attachment, as well as increasing health expenditures. Due to long-term feeding tube use; Infection, leakage, delay in wound healing, trauma caused by repeated placement, as well as oral reluctance are observed. In asphyxia infants, in whom oral-motor dysfunction is common, the transition to oral feeding takes a long time and tube feeding support is required. The effect of hypothermia, which is a general therapeutic intervention that reduces the risk of mortality and morbidity in infants with asphyxia, on oral feeding has been previously studied and shown to have a positive effect. They also found that MR imaging in infants with asphyxia and the need for gastrostomy and tube feeding in those with brainstem involvement were associated.

Various interventions that affect the transition to oral nutrition positively and shorten the discharge time are included in the literature. Stimulation of non-nutritive sucking (NNS) is the most frequently preferred method among these interventions. It has been shown in studies that there are no short-term negative effects of NNS stimulation with the help of a pacifier or gloved finger, and some clinical benefits such as better bottle feeding performance, acceleration of discharge and transition to oral feeding.

The effect of the NNS stimulation method, which has been shown to be effective in preterm infants with large-scale randomized controlled studies, is not known exactly.

The aim of this study is to examine the effect of NNS stimulation applied to oral feeding, feeding skills, weight gain and discharge in asphyxia infants receiving hypothermia treatment.

DETAILED DESCRIPTION:
Perinatal asphyxia is the interruption of fetal blood flow or gas exchange during the perinatal period. Injury to the brain as a result of systemic hypoxia caused by disruption of gas exchange and slowing of cerebral blood flow is called hypoxic ischemic encephalopathy (HIE). Perinatal asphyxia may be maternally related or may occur as a result of conditions related to the placenta and the newborn itself. It may have etiologies such as maternal diseases such as diabetes, hypertension or preeclampsia, uterine rupture, cord compression, congenital airway anomalies of the newborn, neurological disorder, and severe cardiopulmonary disease. According to the World Health Organization (WHO) report, perinatal asphyxia causes 4 million newborn deaths every year and constitutes 23% of total neonatal deaths. Asphyxia, which has effects such as death, seizures and HIE in the short term, has effects such as motor disorders such as cerebral palsy, sensory disorders such as vision and hearing loss, cognitive, neurodevelopmental, behavioral and emotional disorders in the long term. Malnutrition is a problem that can occur both in the short and long term. In the short term, it may have consequences such as orogastric or nasogastric tube feeding due to sucking and/or swallowing dysfunction, prolonged feeding times in the long term, frequent coughing, aspiration pneumonia and gastrostomy. The transition period to full oral feeding in infants with perinatal asphyxia is important in predicting long-term outcomes. The transition to independent oral feeding is accepted as a discharge criterion by the American Academy of Pediatrics, and the long transition from tube feeding to oral feeding prolongs the discharge process. Prolonged transition to oral feeding increases maternal stress as it delays gastrointestinal problems, mother-infant interaction and attachment, as well as increasing health expenditures. Due to long-term feeding tube use; Infection, leakage, delay in wound healing, trauma caused by repeated placement, as well as oral reluctance are observed. In asphyxia infants, in whom oral-motor dysfunction is common, the transition to oral feeding takes a long time and tube feeding support is required. The effect of hypothermia, which is a general therapeutic intervention that reduces the risk of mortality and morbidity in infants with asphyxia, on oral feeding has been previously studied and shown to have a positive effect. They also found that MR imaging in infants with asphyxia and the need for gastrostomy and tube feeding in those with brainstem involvement were associated.

Various interventions that affect the transition to oral nutrition positively and shorten the discharge time are included in the literature. Stimulation of non-nutritive sucking (NNS) is the most frequently preferred method among these interventions. It has been shown in studies that there are no short-term negative effects of NNS stimulation with the help of a pacifier or gloved finger, and some clinical benefits such as better bottle feeding performance, acceleration of discharge and transition to oral feeding.

The effect of the NNS stimulation method, which has been shown to be effective in preterm infants with large-scale randomized controlled studies, is not known exactly. The NNS stimulation method applied in a newborn with severe asphyxia with medical complications was investigated in a case study and it was pointed out that it could have positive results, but more research should be done in this patient group.

The aim of this study is to examine the effect of NNS stimulation applied to oral feeding, feeding skills, weight gain and discharge in asphyxia infants receiving hypothermia treatment.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed with asphyxia,
* to have received hypothermia treatment,
* to have started enteral nutrition,
* to have physiological stability to tolerate NNS stimulation.

Exclusion Criteria:

* Having a craniofacial anomaly,
* having a congenital anomaly,
* being referred to another center/hospital during treatment.

Ages: 34 Months to 41 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Early Feeding Skills Assessment Tool | 1 month
  are the scores obtained by the clinician from the early feeding assessment tool. The minimum score that can be obtained from the scale is 19, and the maximum score is 57. A higher score indicates better feeding skills.
Time from tube feeding to oral intake | 20 days
  how many days the baby transitions from tube feeding to oral intake

SECONDARY OUTCOMES:
discharge time | 1 month
  how many days the baby is discharged from the neonatal intensive care unit
weight gain | 1 month
  is the weight information of the baby at certain intervals

CONTACTS AND LOCATIONS:
Overall Officials: Seyhun Topbas, Study Chair — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harding C, Frank L, Dungu C, Colton N. The use of nonnutritive sucking to facilitate oral feeding in a term infant: a single case study. J Pediatr Nurs. 2012 Dec;27(6):700-6. doi: 10.1016/j.pedn.2012.01.006. Epub 2012 Feb 22. PMID 22366642